CLINICAL TRIAL: NCT04733924
Title: Efficacy and Tolerability of Sensoril® in Improving Immunity and Thereby Reducing Incidence of Upper Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NT/200803/SENSORIL/URT
Record Dates: First submitted 2021-01-21; First posted 2021-02-02 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Immune Health
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Withania somnifera 125 mg (Active Comparator): One capsule before breakfast for 84 days
  Interventions: Other: Aqueous extract of roots plus leaves of Withania somnifera 125 mg
- Withania somnifera 250 mg (Active Comparator): One capsule before breakfast for 84 days
  Interventions: Other: Aqueous extract of roots plus leaves of Withania somnifera 250 mg
- Microcrystalline Cellulose (Placebo Comparator): One capsule before breakfast for 84 days
  Interventions: Other: Microcrystalline Cellulose

INTERVENTIONS:
Other: Aqueous extract of roots plus leaves of Withania somnifera 125 mg — One capsule before breakfast for 84 days
  Arms: Withania somnifera 125 mg
Other: Aqueous extract of roots plus leaves of Withania somnifera 250 mg — One capsule before breakfast for 84 days
  Arms: Withania somnifera 250 mg
Other: Microcrystalline Cellulose — One capsule before breakfast for 84 days
  Arms: Microcrystalline Cellulose

SUMMARY:
to assess the efficacy and safety of a standardized Withania somnifera extract (Sensoril®) as an immunomodulator in individuals suffering from recurrent URTIs. The study population will be administered with this unique blend of WS extract for 12 weeks and will be assessed as per the study designated efficacy and safety variables.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 to ≤ 50 years.
2. High susceptibility to URTIs, defined as ≥ 4 URTI episodes within 12 months.
3. Presence of an active URTI episode (Defined as a score of ≥5 for atleast 2 of following 6 symptoms: runny nose, plugged nose, sneezing, sore throat, scratchy throat, or cough on the WURSS-21 assessment), with onset of symptoms within 48 hours prior to screening.
4. SpO2 ≥ 96% as assessed by fingertip pulse oximetry
5. Commitment to adhere to former diet and physical activities throughout the study period. 6. Able to comply and perform the procedures requested by the protocol (consumption of study medications, filling daily eDiary for health updates, biological sample collection procedures and study visit schedule) 7. Participants who are literate enough to understand the essence of study, are informed about the purpose of the study, and understand their rights. 8. Participants who are able to give written informed consent and are willing to participate in the study.

Exclusion Criteria:

1. History of rhinitis medicamentosa, anatomical nasal obstruction or deformity, nasal reconstructive surgery, etc.
2. Clinical signs or Symptoms indicating lower respiratory tract infection.
3. Known sensitivity to the investigational product or any excipients of the drug product.
4. Any clinically significant abnormalities of the upper respiratory tract (such as stridor, laryngomalacia, etc.)
5. Any clinically significant acute or chronic respiratory illness (such as Sinusitis, pharyngitis/tonsillitis, etc.)
6. Chronic cough of any origin not accompanied to other symptoms of URTI
7. Unable to abstain from any home-based remedies for common cold such as steam inhalation, decoctions, vapour rub, etc. throughout the study period.
8. Presence of uncontrolled type 2 diabetes (Indicated by fasting blood glucose (FBG) ≥126 mg/dL)
9. Presence of uncontrolled hypertension (Defined as Systolic Blood Pressure (SBP) ≥ 140 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 90 mm Hg).
10. Participants with abnormal liver and kidney function tests, defined as:

    * Serum aspartate aminotransferase (AST) and alanine transaminase (ALT) levels > 1.5 × upper level of normal
    * Serum alkaline phosphatase (ALP) levels > 1.5 × upper level of normal
    * Serum creatinine levels > 1.5 × upper level of normal
11. Unable to abstain from ginger, avocado, soy or other known dietary supplements for common cold throughout the study period.
12. Vaccination against influenza or swine flu within 3 months prior to screening.
13. Those who have taken or will be taking or are taking antibiotics, antivirals, steroids, nasal decongestants, antihistamines, or other medications that are expected to alleviate cold symptoms within two weeks prior to randomization.
14. History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's end points.
15. Individuals having a history (in past 2 years) of smoking or currently smoking or using any form of smokeless tobacco.
16. Participation in other clinical trials in last 90 days prior to screening
17. Participants with heavy alcohol consumption, defined as

    * For men: More than 14 standard alcoholic drink (SAD)/week or more than 4 SAD in a day.
    * For women: More than 7 SAD/week or more than 3 SAD in a day. (NOTE - A standard alcoholic drink contains approximately 14 grams of alcohol, which is equivalent to 12 ounces of beer (~5% alcohol), 8.5 ounces of malt liquor (~9% alcohol), 5 ounces of wine (~12% alcohol), 3.5 ounces of fortified wine (e.g., sherry or port), or 1.5 ounces of liquor (distilled spirits; ~40% alcohol).
18. Binge drinkers, defined as 4 or more SAD for women, and 5 or more SAD for men, in a 2-hour time frame.
19. History or presence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
20. Participants who have clinically significant following severe illness (i.e., Cardiovascular, endocrine system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, neuropsychiatric, musculoskeletal, inflammatory, blood and tumors, gastrointestinal diseases, etc.)
21. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
22. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Wisconsin Upper Respiratory Symptom Survey-21 | screening to day 0 and day 57 to day 84
  the effect of IP consumption on incidence of upper respiratory tract infection (URTI) episodes till day 28, 56, and 85 in comparison to placebo as assessed by Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21).

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Dr. Rajesh Kewalramani Clinic, Mumbai, Maharashtra
  - Sanjivani Day Care and Ayurved Center,, Pālghar, Maharashtra
  - Care N Cure Multispeciality Hospital, Thane, Maharashtra